CLINICAL TRIAL: NCT04163536
Title: Comparison of Corticosteroids Versus Placebo on Duration of Ventilatory Support During Severe Acute Exacerbations of COPD Patients in the Intensive Care Unit: a Multicentre Randomized Controlled Trial
Brief Title: Comparison of Corticosteroids vs Placebo on Duration of Ventilatory Support During Severe Acute Exacerbations of COPD Patients in the ICU
Acronym: Corticop
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Alexis FERRE, coordinating investigator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P17/15_corticop
Record Dates: First submitted 2019-10-29; First posted 2019-11-14 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cortisteroids arm (Active Comparator)
  Interventions: Drug: Methylprednisolone
- placebo arm (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Methylprednisolone — In the experimental group, methylprednisolone will be administered intravenously for 5 days at a dose of 1 mg/kg/day. Methylprednisolone will be provided for reconstitution and dilution in 50 ml of NaCl 0.9% solution and administered over 15 minutes, once a day.
  Arms: cortisteroids arm
Drug: Placebos — in the control group, placebo will be administered intravenously for 5 days. Placebo will be identical (color and aspect) to experimental substance, will be provide as a 50 mL of NaCl 0.9% solution and administered intravenously over 15 minutes, once a day.
  Arms: placebo arm

SUMMARY:
The main objective of this study is to determine if the systemic (intravenous) administration of corticosteroids, as compared to placebo, increases the number of ventilator-free days (VFD) and alive at day 28 in COPD patients admitted to an ICU, a step-up unit or a respiratory care unit for an ACRF requiring ventilatory support, either invasive or non-invasive.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 40 years
2. Strongly suspected or documented COPD, defined by the presence of the following criterias:

   * Persistent respiratory symptoms (dyspnoea, chronic cough or sputum)
   * History of exposure to a risk factor such as tobacco smoke
   * If available, pulmonary function tests showing airflow limitation not fully reversible (post-bronchodilator ratio of FEV1/ FVC ratio < 0.7)
3. ACRF, defined by the presence of the two following criteria:

   * COPD exacerbation defined by a change in the patient baseline respiratory symptoms at least 24 hours and requiring a change in regular respiratory medication
   * Acute respiratory failure <24h (polypnea ≥ 30 breaths.min-1 or use of accessory respiratory muscles) requiring ventilatory support, either invasive (implemented because of respiratory distress) or NIV (implemented because of hypercapnic acidosis with PaCO2 ≥ 45 mmHg and pH ≤ 7.35).
4. Admission to an ICU, a step-up unit or a respiratory care unit
5. Inform consent from the patient or his surrogates. In patients who are not able to consent on admission an emergency inclusion procedure will be allowed, with a mandatory delayed consent.
6. Affiliation to (or benefit from) French health insurance system

Exclusion Criteria:

* Previous diagnostic of asthma, according to "GINA" international guidelines (40)
* Recent use of systemic corticosteroids, defined by systemic corticosteroids use in the past 7 days
* Contra-indication of systemic corticosteroids treatment: allergy to corticosteroids, uncontrolled severe arterial hypertension, uncontrolled diabetes mellitus, gastro-intestinal ulcer bleeding
* Pneumothorax at randomization
* Extracorporeal life support (ECMO or ECCO2R) at inclusion
* Moribund patient life expectancy < 3 months
* Pregnancy
* Patients protected by law
* Exclusion period due to other interventional clinical trial enrolment which can influence primary outcome
* Previous inclusion in the present study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the number of ventilator-free days (VFD) and alive at day 28. | day 28
  To determine if the systemic administration of corticosteroids, as compared to placebo, increases the number of ventilator-free days (VFD) and alive at day 28 in COPD patients admitted to an ICU, a step-up unit or a respiratory care unit for an ACRF requiring ventilatory support, either invasive or non-invasive.

SECONDARY OUTCOMES:
NIV failure rate | day 7
  NIV failure rate, defined by intubation within day 7
Duration of NIV and of invasive mechanical ventilation | at day 90
  Duration of Non Invasive Ventilation and of invasive mechanical ventilation
Circulatory and renal support-free days and alive at day 28 | at day 28
  Circulatory and renal support-free days and alive at day 28
Severe hyperglycemia requiring intravenous insulin during the five first days | during the five first days
  Severe hyperglycemia requiring intravenous insulin during the five first days
Gastro-intestinal bleeding | between inclusion and day 28
  acute loss of 2 g/dL of hemoglobin requiring red blood cell transfusion or gastroscopic evaluation
Uncontrolled arterial hypertension | between inclusion and day 28
  unusual hypertension requiring to introduce/add antihypertensive medication (compared to usual medications)
ICU acquired weakness (MRC-score < 48/60) assessed on day 28 or at the time of ICU discharge | at day 28
  Intensive Care Unit acquired weakness (MRC-score < 48/60) assessed on day 28 or at the time of ICU discharge
ICU-acquired infections (especially Ventilator-Associated Pneumonia) | at the time of ICU discharge or day 90
  Intensive Care Unit -acquired infections (especially Ventilator-Associated Pneumonia)
Length of ICU and hospital stay | at day 90
  Length of ICU and hospital stay
ICU and hospital mortality | between inclusion and day 28 or day 90
  ICU and hospital mortality
Day 28 and Day 90 mortality | at Day 28 and Day 90
  Day 28 and Day 90 mortality
Standardized mortality ratio (SMR) | between inclusion and day 90
  Standardized mortality ratio (SMR)
Number of new exacerbation(s)/hospitalization(s) between hospital discharge and Day 90 | at day 90
  Number of new exacerbation(s)/hospitalization(s) between hospital discharge and Day 90
Dyspnea (patient reported outcome) at Day 90 evaluated by clinical assessment test and dyspnea mMRC score | at day 90
  Dyspnea (patient reported outcome) at Day 90 evaluated by clinical assessment test and dyspnea mMRC score
respiratory comfort (patient reported outcome) at Day 90 evaluated by clinical assessment test and dyspnea mMRC score | at day 90
  respiratory comfort (patient reported outcome) at Day 90 evaluated by clinical assessment test and dyspnea mMRC score

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - André Mignot Hospital, Intensive care unit, Le Chesnay, Les Yvelines
  - CHU Angers, Angers
  - CH métropole savoie, Chambéry
  - CHU Louis Mourier, Colombes
  - CHU Henri mondor, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU lille, Lille
  - CHU Lyon, Lyon
  - CH d'Annecy Genevois, Metz-Tessy
  - CHU Nantes, Nantes
  - CHR orléans, Orléans
  - CHU Cochin, Paris
  - Hôpital européen Georges pompidou, Paris
  - Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - Hopital Foch, Suresnes
  - CHRU Tours, Tours